CLINICAL TRIAL: NCT04246437
Title: [18F]F-DOPA Imaging in Patients With Autonomic Failure
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Claassen (Other)
Responsible Party: Sponsor-Investigator, Daniel Claassen, Professor of Neurology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 192021
Record Dates: First submitted 2020-01-25; First posted 2020-01-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Autonomic Failure; Pure Autonomic Failure; Parkinson Disease; Multiple System Atrophy; Dementia With Lewy Bodies
Keywords: FDOPA; PET
MeSH Terms: conditions — Pure Autonomic Failure; Parkinson Disease; Multiple System Atrophy; Lewy Body Disease | interventions — fluorodopa F 18; Carbidopa; entacapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]F-DOPA (Experimental): All patients will receive [18F]F-DOPA for PET imaging to measure pre-synaptic dopamine in the brain.
  Interventions: Drug: [18F]FDOPA; Drug: Carbidopa 200mg oral dose; Drug: Entacapone 400mg oral dose

INTERVENTIONS:
Drug: [18F]FDOPA — Patients will receive a 3-D emission scan following a 6-8 mCi slow bolus injection of [18F]FDOPA over a 30 second period. Serial scans are started simultaneously with the bolus injection of radiotracer and are obtained for approximately 95 minutes.
Drug: Carbidopa 200mg oral dose — 30 minutes prior to the PET scan, patients will receive the 200mg oral dose of carbidopa to prevent peripheral [18F]FDOPA metabolism to increase signal-to-noise ratio of the imaging.
  Other Names: Lodosyn
Drug: Entacapone 400mg oral dose — 30 minutes prior to the PET scan, patients will receive the 400mg oral dose of entacapone to prevent peripheral [18F]FDOPA metabolism to increase signal-to-noise ratio of the imaging.
  Other Names: Comtan

SUMMARY:
Alpha-synucleinopathies refer to age-related neurodegenerative and dementing disorders, characterized by the accumulation of alpha-synuclein in neurons and/or glia. The anatomical location of alpha-synuclein inclusions (Lewy Bodies) and the pattern of progressive neuronal death (e.g. caudal to rostral brainstem) give rise to distinct neurological phenotypes, including Parkinson's disease (PD), Multiple System Atrophy (MSA), Dementia with Lewy Bodies (DLB). Common to these disorders are the involvement of the central and peripheral autonomic nervous system, where Pure Autonomic Failure (PAF) is thought (a) to be restricted to the peripheral autonomic system, and (b) a clinical risk factor for the development of a central synucleinopathy, and (c) an ideal model to assess biomarkers that predict phenoconversion to PD, MSA, or DLB. Such biomarkers would aid in clinical trial inclusion criteria to ensure assessments of disease- modifying strategies to, delay, or halt, the neurodegenerative process. One of these biomarkers may be related to the neurotransmitter dopamine (DA) and related changes in the substantia nigra (SN) and brainstem. [18F]F-DOPA is a radiolabeled substrate for aromatic amino acid decarboxylase (AAADC), an enzyme involved in the production of dopamine. Use of this radiolabeled substrate in positron emission tomography (PET) may provide insight to changes in monoamine production and how they relate to specific phenoconversions in PAF patients. Overall, this study aims to identify changes in dopamine production in key regions including the SN, locus coeruleus, and brainstem to distinguish between patients with PD, MSA, and DLB, which may provide vital information to predict conversion from peripheral to central nervous system disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis if pure autonomic failure
2. Patients with autonomic failure and possible PD, MSA, or DLB
3. Healthy adults aged 18 and above
4. Clinical exam confirming clinical designation

Exclusion Criteria:

* Subjects who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.), because such devices may be displaced or malfunction.
* Subjects who have any type of ferromagnetic bioimplant that could potentially be displaced.
* Subjects who have cerebral aneurysm clips.
* Subjects who may have shrapnel imbedded in their bodies (such as from war wounds), metal workers and machinists (potential for metallic fragments in or near the eyes).
* Subjects who are pregnant, because the effects of high field MRI on fetuses are not yet known.
* Minors (younger than 18 years)

Also excluded are subjects incapable of giving informed written consent:

* Subjects who cannot adhere to the experimental protocols for any reason, or have an inability to communicate with the researcher.
* Subjects who have limited mental ability to give informed consent, mentally retarded, altered mental status, mental disability, confusion, or psychiatric disorders.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Differences in FDOPA uptake across patient populations | 95 minutes post-PET after start of PET imaging
  Specific FDOPA uptake, Ki, will be calculated via a reference Logan plot to provide voxelwise measurements of FDOPA uptake. Mean uptake will be assessed in brain regions-of-interest in 40 participants to assess potential differences across different autonomic failure-related diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States